CLINICAL TRIAL: NCT07216859
Title: Screening Cardiometabolic Opportunities Using Transformative Echocardiography Artificial Intelligence (SCOUT Echo-AI)
Acronym: SCOUT Echo-AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Stanford University (Other); Massachusetts General Hospital (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Ouyang, Int Med-Cardio Non-Invasive, Kaiser Permanente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2356334; 25AHAAI1487693 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI Notification (EchoNet-Liver-Flagged patients) (Experimental): Participants whose prior transthoracic echocardiograms are flagged by an AI model (EchoNet-Liver) as high risk for MASLD and/or cirrhosis, a notification is delivered to the primary treating clinician, or undergoes a structured diagnostic workflow.
  Interventions: Other: AI-Enabled Identification (EchoNet-Liver)

INTERVENTIONS:
Other: AI-Enabled Identification (EchoNet-Liver) — AI-generated notifications to clinicians about possible undiagnosed liver disease (MASLD and/or Cirrhosis) detected from Transthoracic Echocardiogram

SUMMARY:
The goal of this prospective, multicenter, open-label, blinded end-point pragmatic study is to evaluate an artificial intelligence (AI)-augmented echocardiography screening approach for early detection of metabolic dysfunction associated steatotic liver disease (MASLD) and/or cirrhosis, in patients undergoing routine transthoracic echocardiograms (TTEs).

The main question it aims to answer is to:

1. Evaluate notification responsiveness and rates of confirmatory testing for patients identified as high risk for having liver disease to determine whether optimized notifications increase timely confirmatory testing and treatment initiation versus standard of care assessment.
2. Compare time to diagnosis, treatment uptake, and clinical outcomes (hospitalizations, incident ASCVD, mortality) between cohorts identified as high risk by the AI algorithm and comparison groups to determine whether AI guided screening shortens time to diagnosis and increases appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Underwent routine TTE within site defined recent timeframe and flagged as high risk for MASLD and/or cirrhosis by the AI model using pre specified threshold.
* Able to provide informed consent; reachable for follow up.

Exclusion Criteria:

* Inability to consent or communicate.
* Enrollment in hospice or life expectancy so limited that additional evaluation would not be appropriate per clinician judgment.
* Clinical circumstances where immediate alternative diagnostic pathways supersede study procedures (e.g., acute decompensation requiring urgent management).
* Prior liver or kidney transplant.
* Patient unwilling to undergo prospective testing for liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) of the AI algorithm for detecting MASLD and/or cirrhosis confirmed within 12 months of AI identification. | From enrollment to end of follow up at 1 year.
  Numerator: Participants with clinician-confirmed diagnosis of later stage MASLD and/or cirrhosis after confirmatory evaluation.
  Denominator:
  * Participants with positive AI screen who were enrolled and evaluated.
  * The intervention is the clinician referral or referral testing workflow. The clinicians ultimately have discretion to avoid further downstream testing if pretest probability is felt to be too low. If a clinician determines no further testing is warranted despite high risk assessment by AI, the participant will be classified as a false positive (still counted in the denominator).

SECONDARY OUTCOMES:
Time to diagnosis of MASLD/cirrhosis | Followed up to 24 months post notification.
  Time (days) from AI identification to first confirmatory diagnosis
Time to diagnosis for MASLD with F2 fibrosis or greater | Followed up to 24 months post notification.
  Time (days) from AI identification to first confirmatory diagnosis
Time to diagnosis for steatotic liver disease | Followed up to 24 months post notification.
  Time (days) from AI identification to first confirmatory diagnosis
Time to confirmatory imaging | Followed up to 24 months post notification.
  Time (days) from AI identification
Time to initiation of targeted treatment | Followed up to 24 months post notification.
  Time (days) from AI identification
All-cause mortality | Followed up to 24 months post notification.
  Time (days) from AI identification
All-cause hospitalization | Followed up to 24 months post notification.
  Time (days) from AI identification
Heart failure hospitalization | Followed up to 24 months post notification.
  Time (days) from AI identification (Defined as admission with IV diuretics or elevated BNP)
Cardiovascular hospitalization | Followed up to 24 months post notification.
  Time (days) from AI identification for Cardiovascular hospitalization (defined by principal ICD9/10 code)
Hepatic decompensation hospitalization | Followed up to 24 months post notification.
  Time (days) from AI identification for hepatic decompensation hospitalization (defined by ascites, hepatic encephalopathy, variceal bleeding, hepatocellular carcinoma, or liver transplantation)
New ASCVD diagnosis | Followed up to 24 months post notification.
  Time (days) from AI identification

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Healthcare, Palo Alto, California
  - Kaiser Permanente, Pleasanton, California
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided